CLINICAL TRIAL: NCT04273139
Title: Phase II Study on the Combination of Ibrutinib and Venetoclax in Treatment naïve Patients With Waldenström Macroglobulinemia
Brief Title: Ibrutinib + Venetoclax in Untreated WM
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: AbbVie (Industry); Pharmacyclics LLC. (Industry)
Responsible Party: Principal Investigator, Jorge J. Castillo, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 19-651
Record Dates: First submitted 2020-02-14; First posted 2020-02-17 (Actual); Results first posted 2024-04-23 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Waldenstrom Macroglobulinemia; MYD88 Gene Mutation
Keywords: Waldenstrom Macroglobulinemia; ibrutinib; venetoclax
MeSH Terms: conditions — Waldenstrom Macroglobulinemia | interventions — ibrutinib; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ibrutinib and Venetoclax (Experimental): The research study procedures include screening for eligibility and study treatment including evaluations and follow up visits.
  * Ibrutinib will be administered at a predetermined dose, once daily for 28 days
  * TLS Prophylaxis (Treatment to reduce risk of tumor lysis syndrome) prior to first dose of venetoclax (and for at least the first 2 weeks of treatment)
  * Venetoclax Cycle 2-24. PO daily, predetermined dosage ramp up during cycle 2.
  Interventions: Drug: IBRUTINIB; Drug: Venetoclax

INTERVENTIONS:
Drug: IBRUTINIB — Ibrutinib Cycle 1-24 will be administered at a predetermined dose, once daily for 28 days
  Other Names: Imbruvica
Drug: Venetoclax — Venetoclax Cycle 2-24 will be administered daily for 28 days. Predetermined dosage ramp up schedule during cycle 2.
  Other Names: Venclexta

SUMMARY:
This study evaluates the safety and efficacy of Ibrutinib combined with Venetoclax (IVEN) in the treatment of adults diagnosed with Waldenstrom's macroglobulinemia (WM) cancer with a specific MYD88 gene mutation.

This research study involves an experimental drug combination of targeted therapies.

The names of the study drugs involved in this study are:

* Venetoclax
* ibrutinib

DETAILED DESCRIPTION:
* This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational drug to learn whether the drug works in treating a specific disease. "Investigational" means that the drug is being studied.
* The names of the study drugs involved in this study are:

  * Venetoclax
  * ibrutinib
* The research study procedures include screening for eligibility and study treatment including evaluations and follow up visits.

  * Participants will be on the research study for up to 2 years on combined venetoclax and ibrutinib and 4 years of follow-up .
  * It is expected that about 50 people will take part in this research study.
* The U.S. Food and Drug Administration (FDA) has not approved venetoclax for your specific disease but it has been approved for other uses.

  -- Venetoclax is a targeted therapy that blocks BCL-2, a protein that is important for the survival of WM cells. Laboratory studies and early clinical data have shown that the investigational new agent, venetoclax, may kill cancer cells and may cause tumors to shrink.
* The U.S. Food and Drug Administration (FDA) has approved ibrutinib as a treatment option for this disease.

  --Ibrutinib is a targeted therapy that blocks BTK. It has been FDA approved in chronic lymphocytic leukemia (CLL), small lymphocytic lymphoma (SLL), mantle cell lymphoma (MCL), marginal zone lymphoma (MZL), chronic graft vs. host disease (cGVHD), and Waldenstrom's macroglobulinemia (WM). It is also used in research studies in participants with recurrent B-cell lymphoma), diffuse large B-cell lymphoma (DLBCL), and prolymphocytic leukemia. In a study of ibrutinib in relapsed/refractory WM patients, response rates were high and the treatment was well tolerated.
* The U.S. Food and Drug Administration (FDA) has not approved the combination of ibrutinib and venetoclax as a treatment for any disease.
* The U.S. Food and Drug Administration (FDA) has not approved the MYD88 test. This test is investigational.

ELIGIBILITY:
Inclusion Criteria:

* Participants must meet the following criteria on screening examination to be eligible to participate. Screening evaluations including consent, physical exam, and laboratory assessments will be done within 30 days prior to Cycle 1 Day 1. Bone marrow biopsy & aspirate, and CT C/A/P will be done within 90 days prior to Cycle 1 Day 1.
* Clinicopathological diagnosis of Waldenström macroglobulinemia [28].
* Known tumor expression of mutated MYD88 performed by a CLIA certified laboratory.
* Symptomatic disease meeting criteria for treatment using consensus panel criteria from the Second International Workshop on Waldenström macroglobulinemia [29].
* Participants with symptomatic hyperviscosity (e.g. nosebleeds, headaches, blurred vision) must undergo plasmapheresis prior to treatment initiation.
* Age ≥ 18 years
* ECOG performance status ≤2 (see Appendix A)
* Measurable disease, defined as presence of serum immunoglobin M (IgM) with a minimum IgM level of >2 times the upper limit of normal of each institution is required
* At the time of screening, participants must have acceptable organ and marrow function as defined below:

  * Absolute neutrophil count ≥500/uL (no growth factor permitted)
  * Platelets ≥50,000/uL (no platelet transfusions permitted)
  * Hemoglobin ≥ 7 g/dL (transfusions permitted)
  * Total bilirubin < 1.5 x institutional ULN
  * AST(SGOT)/ALT(SGPT) ≤2.5 × institutional ULN
  * Estimated GFR ≥30 mL/min
* Females of childbearing potential (FCBP) must use one reliable form of contraception or have complete abstinence from heterosexual intercourse during the following time periods related to this study: 1) while participating in the study; and 2) for at least 90 days after discontinuation from the study. FCBP must be referred to a qualified provider of contraceptive methods if needed. FCBP must have a negative serum pregnancy test at screening.
* Men must agree to use a latex condom during treatment and for up to 90 days after the last dose of ibrutinib or venetoclax during sexual contact with a FCBP
* Ability to understand and the willingness to sign a written informed consent document.
* Exclusion Criteria
* Participants who exhibit any of the following conditions at screening will not be eligible for admission into the study:
* Participants who have one or more prior systemic therapies for WM.
* Participants who are receiving any other investigational agents.
* Participants with known CNS lymphoma.
* Participants with known history of Human Immunodeficiency Virus (HIV), chronic hepatitis B virus (HBV) or hepatitis C (HCV) requiring active treatment. Note: Participants with serologic evidence of prior vaccination to HBV (i.e., HBs Ag-, and anti-HBs+ and anti-HBC-) and positive anti-HBc from IVIG may participate.
* Concurrent administration of medications or foods that are moderate or strong inhibitors or inducers of CYP3A within 7 days prior to first dose of study drug.
* Participants with chronic liver disease and hepatic impairment meeting Child-Pugh class C (Appendix B).
* Concurrent administration of warfarin.
* Concurrent systemic immunosuppressant therapy within 21 days of the first dose of study drug.
* Vaccinated with live, attenuated vaccines within 4 weeks of first dose of study drug.
* Recent infection requiring systemic treatment that was completed ≤ 14 days before the first dose of the study drug.
* Known bleeding disorders (e.g., congenital von Willebrand's disease or hemophilia)
* History of stroke or intracranial hemorrhage within 6 months prior to enrollment.
* Major surgery within 4 weeks of first dose of study drug.
* Malabsorption syndrome or other condition that precludes enteral route of administration.
* Female participants who are pregnant, breastfeeding, or planning to become pregnant while enrolled in this study or within 90 days of last dose of study drug.
* Male participants who plan to father a child while enrolled in this study or within 90 days after the last dose of study drug
* Participants with known history of alcohol or drug abuse.
* Participants with inability to swallow pills.
* On any active therapy for other malignancies with the exception of topical therapies for basal cell or squamous cell cancers of the skin.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Participants with a history of non-compliance to medical regimens.
* Participants who are unwilling or unable to comply with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2020-07-09 (Actual); Primary Completion 2022-06-06 (Actual); Study Completion 2028-02-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Jorge J Castillo, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu

REFERENCES:
- [Derived] Castillo JJ, Branagan AR, Sermer D, Flynn CA, Meid K, Little M, Stockman K, White T, Canning A, Guerrera ML, Kofides A, Liu S, Liu X, Richardson K, Tsakmaklis N, Patterson CJ, Hunter ZR, Treon SP, Sarosiek S. Ibrutinib and venetoclax as primary therapy in symptomatic, treatment-naive Waldenstrom macroglobulinemia. Blood. 2024 Feb 15;143(7):582-591. doi: 10.1182/blood.2023022420. PMID 37971194

RESULTS

PARTICIPANT FLOW:
Groups:
- Ibrutinib and Venetoclax: The research study procedures include screening for eligibility and study treatment including evaluations and follow up visits.
  * Ibrutinib will be administered at a predetermined dose, once daily for 28 days
  * TLS Prophylaxis (Treatment to reduce risk of tumor lysis syndrome) prior to first dose of venetoclax (and for at least the first 2 weeks of treatment)
  * Venetoclax Cycle 2-24. PO daily, predetermined dosage ramp up during cycle 2.
  IBRUTINIB: Ibrutinib Cycle 1-24 will be administered at a predetermined dose, once daily for 28 days
  Venetoclax: Venetoclax Cycle 2-24 will be administered daily for 28 days. Predetermined dosage ramp up schedule during cycle 2.
Period: Overall Study
Arm/Group | Ibrutinib and Venetoclax
Started | 45
Completed | 45
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Ibrutinib and Venetoclax
Number analyzed (Participants) | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 25
Age, Continuous [Median (Full Range); unit: years] | 67 [39 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 43
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 42
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 45

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Very Good Partial Response Within 24 Cycles of Therapy
Description: Proportion of patients with VGPR to therapy within 24 cycles of therapy initiation. (VGPR is >90% reduction in serum IgM from baseline)
Time Frame: The primary objective of VGPR within 24 cycles of therapy was assessed starting at Cycle 3 Day 1 through the End of Treatment visit, range of 2 to 21 months after the initiation of therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | Ibrutinib and Venetoclax
Number analyzed (Participants) | 45
Participants | 19

2. Secondary Outcome: Number of Participants With Complete Response (CR) After 6 Cycles
Description: Proportion of patients with a complete response after 6 cycles of therapy. A complete response (CR) is defined as having resolution of WM related symptoms, normalization of serum IgM levels with complete disappearance of IgM paraprotein by immunofixation, and resolution of any adenopathy or splenomegaly.
Time Frame: 6 Cycles (28 day cycle)
Measure: Count of Participants; unit: Participants
Arm/Group | Ibrutinib and Venetoclax
Number analyzed (Participants) | 45
Participants | 0

3. Secondary Outcome: Number of Participants With Complete Response (CR) After 12 Cycles
Description: Proportion of patients with a complete response after 12 cycles of therapy. A complete response (CR) is defined as having resolution of WM related symptoms, normalization of serum IgM levels with complete disappearance of IgM paraprotein by immunofixation, and resolution of any adenopathy or splenomegaly.
Time Frame: 12 Cycles (28 day cycle)
Measure: Count of Participants; unit: Participants
Arm/Group | Ibrutinib and Venetoclax
Number analyzed (Participants) | 45
Participants | 0

4. Secondary Outcome: Number of Participants With Complete Response (CR) After 24 Cycles
Description: Proportion of patients with a complete response after 24 cycles of therapy. A complete response (CR) is defined as having resolution of WM related symptoms, normalization of serum IgM levels with complete disappearance of IgM paraprotein by immunofixation, and resolution of any adenopathy or splenomegaly.
Time Frame: Complete response to therapy was assessed starting at Cycle 3 Day 1 through the End of Treatment visit, range of 2 to 21 months after the initiation of therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | Ibrutinib and Venetoclax
Number analyzed (Participants) | 45
Participants | 0

5. Secondary Outcome: Overall Response
Description: Proportion of patients with minor response (MR) , partial response (PR), very good partial response (VGPR), or complete response (CR) to therapy.
Time Frame: 72 months
Reporting Status: Not Posted, anticipated posting 2028-01

6. Secondary Outcome: Rate of VGPR at 30 Months
Description: Proportion of patients with a VGPR at 30 months from beginning therapy.
Time Frame: 30 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Ibrutinib and Venetoclax
Number analyzed (Participants) | 45
Participants | 9

7. Secondary Outcome: Median Time to Response
Description: Time from treatment initiation until achievement of a minor response (reduction in serum IgM >25%) or better.
Time Frame: 24 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ibrutinib and Venetoclax
Number analyzed (Participants) | 45
months | 0.9 [0.9 to 1]

8. Secondary Outcome: Median Time to Major Response
Description: Time from treatment initiation until partial response or better (>50% reduction in serum IgM)
Time Frame: 24 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ibrutinib and Venetoclax
Number analyzed (Participants) | 45
months | 1.8 [1.4 to 1.9]

9. Secondary Outcome: Progression Free Survival (PFS) at 24 Months
Description: Time from initiation of therapy until disease progression (>25% increase in serum IgM and 500 mg/dL absolute increase).
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Ibrutinib and Venetoclax
Number analyzed (Participants) | 45
Participants | 34

10. Secondary Outcome: Progression Free Survival (PFS) at 36 Months
Description: Time from initiation of therapy until disease progression (>25% increase in serum IgM and 500 mg/dL absolute increase).
Time Frame: 36 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Ibrutinib and Venetoclax
Number analyzed (Participants) | 45
Participants | 21

11. Secondary Outcome: Progression Free Survival (PFS) at 48 Months
Description: Time from initiation of therapy until disease progression (>25% increase in serum IgM and 500 mg/dL absolute increase).
Time Frame: 48 Months
Reporting Status: Not Posted, anticipated posting 2026-01

12. Secondary Outcome: Progression Free Survival (PFS) at 60 Months
Description: Time from initiation of therapy until disease progression (>25% increase in serum IgM and 500 mg/dL absolute increase).
Time Frame: 60 Months
Reporting Status: Not Posted, anticipated posting 2027-01

13. Secondary Outcome: Overall Survival
Description: Time from initiation of therapy until death
Time Frame: 72 months
Reporting Status: Not Posted, anticipated posting 2028-01

14. Secondary Outcome: Time to Next Treatment
Description: Time from initiation of IVEN protocol therapy until initiation of new line of therapy.
Time Frame: 72 months
Reporting Status: Not Posted, anticipated posting 2028-01

15. Secondary Outcome: Number of Participants With Treatment Related Adverse Events as Assessed (CTCAE) Version 5.0
Description: CTCAE version 5.0
Time Frame: 6 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Ibrutinib and Venetoclax
Number analyzed (Participants) | 45
Participants | 45

ADVERSE EVENTS:
Time Frame: Adverse events were collected from study treatment initiation through 30 days of last dose (e.g. 2 years)
Arm/Group | Ibrutinib and Venetoclax
All-Cause Mortality (participants affected / at risk) | 2/45
Serious Adverse Events (participants affected / at risk) | 10/45
Other Adverse Events (participants affected / at risk) | 45/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ibrutinib and Venetoclax (N=45)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Aspiration pneumonia (Infections and infestations) | 1 (1)
Intracranial hemorrhage (Nervous system disorders) | 1 (1)
Laboratory Tumor Lysis Syndrome (Metabolism and nutrition disorders) | 1 (1)
Hyperphosphatemia (Metabolism and nutrition disorders) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 2 (2)
Cardiac arrest (Cardiac disorders) | 2 (2)
Hematoma (Vascular disorders) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ibrutinib and Venetoclax (N=45)
Anemia (Blood and lymphatic system disorders) | 8 (8)
Easy bleeding (Blood and lymphatic system disorders) | 6 (6)
Petechia (Blood and lymphatic system disorders) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 3 (3)
Chest pain (Cardiac disorders) | 3 (3)
Palpitations (Cardiac disorders) | 9 (9)
Blurred vision (Eye disorders) | 1 (1)
Dry eye (Eye disorders) | 1 (1)
Eye pain (Eye disorders) | 2 (2)
Floaters (Eye disorders) | 1 (1)
Retinal vein occlusion (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 4 (4)
Bloating (Gastrointestinal disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 8 (8)
Diarrhea (Gastrointestinal disorders) | 26 (26)
Dry mouth (Gastrointestinal disorders) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 1 (1)
C. difficile infection (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 7 (7)
Gastroenteritis (Gastrointestinal disorders) | 2 (2)
GERD (Gastrointestinal disorders) | 13 (13)
Increased appetite (Gastrointestinal disorders) | 1 (1)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 16 (16)
Nausea (Gastrointestinal disorders) | 20 (20)
Vomiting (Gastrointestinal disorders) | 2 (2)
Chills (General disorders) | 1 (1)
Edema limbs (General disorders) | 4 (4)
Fatigue (General disorders) | 12 (12)
Fever (General disorders) | 2 (2)
Increased sensitivity to cold (General disorders) | 1 (1)
Generalized edema (General disorders) | 3 (3)
Malaise (General disorders) | 1 (1)
Folliculitis (Infections and infestations) | 2 (2)
Gum infection (Infections and infestations) | 1 (1)
Herpes simplex reactivation (Infections and infestations) | 1 (1)
COVID-19 infection (Infections and infestations) | 5 (5)
Nail infection (Infections and infestations) | 1 (1)
Papulopustular rash (Infections and infestations) | 2 (2)
Shingles (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 2 (2)
Skin infection (Infections and infestations) | 2 (2)
Soft tissue infection (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 4 (4)
Urinary tract infection (Infections and infestations) | 3 (3)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 16 (16)
Fall (Injury, poisoning and procedural complications) | 2 (2)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1)
Wound complication (Injury, poisoning and procedural complications) | 3 (3)
ALT elevation (Investigations) | 3 (3)
Alkaline phosphatase increased (Investigations) | 1 (1)
AST elevation (Investigations) | 2 (2)
LDH increased (Investigations) | 1 (1)
Cardiac troponin t increased (Investigations) | 1 (1)
Creatinine increased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 16 (16)
Platelet count decreased (Investigations) | 6 (6)
Weight gain (Investigations) | 1 (1)
Weight loss (Investigations) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 5 (5)
Hyperphosphatemia (Metabolism and nutrition disorders) | 7 (7)
Hyperuricemia (Metabolism and nutrition disorders) | 2 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Laboratory Tumor Lysis Syndrome (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 (11)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Stiff joints (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle cramps (Musculoskeletal and connective tissue disorders) | 7 (7)
Plantar fascitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 7 (7)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4)
DCIS left breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Dizziness (Nervous system disorders) | 10 (10)
Dysgeusia (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 6 (6)
Imbalance (Nervous system disorders) | 2 (2)
Paresthesia (Nervous system disorders) | 3 (3)
Presyncope (Nervous system disorders) | 2 (2)
Anxiety (Psychiatric disorders) | 1 (1)
Hallucinations (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 3 (3)
Irritability (Psychiatric disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 2 (2)
Urinary frequency (Renal and urinary disorders) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Urinary urgency (Renal and urinary disorders) | 1 (1)
Irregular menstruation (Reproductive system and breast disorders) | 1 (1)
Bleeding (Reproductive system and breast disorders) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8 (8)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 9 (9)
Hair thining (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 (3)
Nail changes (Skin and subcutaneous tissue disorders) | 6 (6)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritis (Skin and subcutaneous tissue disorders) | 2 (2)
Purpura (Skin and subcutaneous tissue disorders) | 3 (3)
Maculopapular Rash (Skin and subcutaneous tissue disorders) | 3 (3)
Fragile skin (Skin and subcutaneous tissue disorders) | 11 (11)
Lesion (Skin and subcutaneous tissue disorders) | 3 (3)
Nodular rash (Skin and subcutaneous tissue disorders) | 1 (1)
Skin changes (Skin and subcutaneous tissue disorders) | 2 (2)
Rash not otherwise specified (Skin and subcutaneous tissue disorders) | 7 (7)
skin induration (Skin and subcutaneous tissue disorders) | 1 (1)
Hot flashes (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 4 (4)
Raynaud's symptoms (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-11): https://cdn.clinicaltrials.gov/large-docs/39/NCT04273139/Prot_SAP_000.pdf